CLINICAL TRIAL: NCT05052021
Title: A Prospective Observational Cohort Study of Patient-reported Outcomes After Surgery Using a Digital Health Platform
Brief Title: The South African Collaborative Surgical Outcomes Study (SACSOS)
Acronym: SACSOS
Status: Not yet recruiting | Type: Observational
Sponsor: Sefako Makgatho Health Sciences University (Other)
Collaborators: Medical Research Council, South Africa (Other); University of Cape Town (Other)
Responsible Party: Principal Investigator, Hyla-Louise Kluyts, Professor, Sefako Makgatho Health Sciences University
Other Study IDs: SMUREC/M/184/2020
Record Dates: First submitted 2021-09-14; First posted 2021-09-22 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Complications
Keywords: Outcome measures; Peri-operative care; Patient-centered care
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients within the private healthcare sector: Patients from private sector hospitals in South Africa accommodating the use of the Bespoke Surgical Institute (BSI) Deep Health clinical data platform.
  Interventions: Other: Public or Private Sector Patients
- Patients within the public healthcare sector.: Patients admitted for surgery at Dr George Mukhari Academic Hospital, Gauteng Department of Health.
  Interventions: Other: Public or Private Sector Patients

INTERVENTIONS:
Other: Public or Private Sector Patients — No intervention will be done. Two groups of patients will be recruited: patients receiving surgery in the Private Healthcare Sector, and patients receiving surgery in the Public Healthcare Sector

SUMMARY:
Improving quality of perioperative care depends on reliable measurement of clinically important and patient-centred data, that will allow collaborative decision-making between patient and clinician. The use of digital health tools to share person-centric data with the aim of improving quality of care is encouraged by the World Health Organization Global Strategy on Digital Health. With virtual and online communication becoming a universal feature of modern life, there is a promising opportunity to engage patients and clinicians in perioperative data collection using digital health platforms. The Perioperative Shared Health Record (PSHR), developed by Safe Surgery South Africa, provides the opportunity to capture standardised patient-centric postoperative outcomes measures, like Quality of Recovery (QOR), Health Related Quality of Life (HRQOL), the WHO Disability Assessment Schedule (WHODAS). These are all standardised measures and questionnaires, which have been recommended by working groups focused on the patient's experience after surgery. The PSHR enables sharing of data between the surgical patient and his/her clinical team (surgeons and anaesthetists).

DETAILED DESCRIPTION:
SACSOS is a patient-centered prospective observational cohort study.

Initially, clinical teams in the South African private health care sector will be approached. In later phases of the study, recruitment will include eligible patients in the South African public health care sector.

Patient engagement and -participation will be sought during the recruitment process by engaging with the clinical team (surgeon, anaesthetist, hospital clinical manager) for individual patient care (at a micro level); in data collection using a patient-centric platform; and in the follow up after surgery. Data will be collected by patients using a digital platform, the Perioperative Shared Health Record (PSHR). De-identified data will be extracted from the database at predetermined intervals and made available to the principal investigator for analysis.

The PSHR will be updated to optimise health information exchange between the surgical patient and clinical team members during the study.

Participation from health care providers will be in a team-based approach, including surgeon(s) and/or anaesthetist(s) at each specific center. A core group of participating centers will be identified.

The study will focus on patient participation with the web-based platform as the primary recruitment method. This will reduce the need for clinician input, and promote greater patient-centeredness. Patient participation and data capturing require internet access to the web-based platform.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients presenting for any surgical procedure at South African hospitals during the specified study period.

Exclusion Criteria:

* Patients unable to provide consent to participation.
* Patients whose legal guardian is unable to provide consent to participation (if applicable).
* Patients unable to nominate next-of-kin, guardian of or a person of their choice, as their representative during follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To enable a patient-centred approach, patients will be invited to participate in the study by a member of the clinical team responsible for their care. Initially, clinical teams in the South African private health care sector will be approached. In later phases of the study, recruitment will include eligible patients in the South African public health care sector.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
To describe the relationship between preoperative and 6-month postoperative health-related quality of life in South African surgical patients. | 6 Months post-operatively
  Health Related Quality of Life, measured with the EQ-5D-5L score, preoperatively and at 6 months postoperatively

SECONDARY OUTCOMES:
To describe the relationship between patient comorbidities, surgical characteristics and postoperative patient- reported outcomes measures (quality of recovery, health-related quality of life). | 24-48 hours postoperatively
  Quality of recovery (QoR) preoperatively and at 24-48 hours postoperatively
To assess data quality (accuracy) of the adapted patient-reported POMS by comparison with completed provider POMS. | 5 days postoperatively
  Amended Postoperative Morbidity Survey (POMS) postoperatively after 5 days
To compare data quality (completeness) for patient-reported outcomes and provider POMS between public and private sector settings. | 5-7 days postoperatively
  POMS recorded by surgeon at discharge from hospital after surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Biccard, PhD, Principal Investigator — University of Cape Town; Hyla-Louise Kluyts, DMed, Principal Investigator — Sefako Makgatho Health Sciences University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Website for Safe Surgery South Africa. Surgery South Africa, a non-profit company (NPC) will act as custodian of data captured using the Perioperative Shared Health Record (PSHR) platform. — https://safesurgery.co.za/

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-05-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT05052021/Prot_SAP_ICF_001.pdf